CLINICAL TRIAL: NCT05850065
Title: Assessment of Gingival Health Following Different Retraction Techniques in Restorative Rubber-Dam Isolation
Brief Title: Assessment of Gingival Health Following Rubber-Dam Isolation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09.2023.126
Record Dates: First submitted 2023-04-05; First posted 2023-05-09 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Gingival Recession, Localized
Keywords: Retraction; Rubber-dam isolation; Clamp; Gingival health
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hu-Friedy 212 clamp (Other): Hu-Friedy 212 clamp will used for the retraction.
  Interventions: Other: Hu-Friedy 212 clamp
- dental floss using the simple knot tie method (Other): Dental floss using the simple knot tie method will used for the retraction.
  Interventions: Other: dental floss using the simple knot tie method
- Using Hu-Friedy 212 clamp and dental floss using the simple knot tie method together (Other): Using Hu-Friedy 212 clamp and dental floss using the simple knot tie method together will used for the retraction.
  Interventions: Other: Hu-Friedy 212 clamp; Other: dental floss using the simple knot tie method
- Coltene B4 clamp (Other): Coltene B4 clamp will used for the retraction.
  Interventions: Other: Coltene B4 clamp

INTERVENTIONS:
Other: Hu-Friedy 212 clamp — Hu-Friedy 212 clamp is normally used for the retraction with rubber-dam
  Arms: Hu-Friedy 212 clamp; Using Hu-Friedy 212 clamp and dental floss using the simple knot tie method together
Other: dental floss using the simple knot tie method — Dental floss using the simple knot tie method is normally used for the retraction with rubber-dam
  Arms: Using Hu-Friedy 212 clamp and dental floss using the simple knot tie method together; dental floss using the simple knot tie method
Other: Coltene B4 clamp — Coltene B4 clamp is normally used for the retraction with rubber-dam
  Arms: Coltene B4 clamp

SUMMARY:
The aim of this study is to evaluate the effect of retraction techniques on gingival health. Four different method (212 clamp (Hu-Friedy, USA); Brinker B4 clamp (Coltene Hygenic, USA); dental floss using the simple knot tie method; and using the simple knot tie and 212 clamp together) will evaluated. After rubber dam isolation restorations will be performed, each restoration will take maximum 30 minutes.

Changes in periodontal tissues will be evaluate; using plaque index, bleeding on probing, probing depth, keratinized gingiva, attached gingiva, relative gingival margin level, relative attachment level and VAS (visual analogue scale) scoring and patient comfort levels after the procedure at different times (pre-restoration, after restoration, 1 week, 1 month, 3 month). The evaluation time is planned not to exceed 10 minutes, restorations are done by a single specialist in Marmara University Restorative Dentistry Department.

DETAILED DESCRIPTION:
In the present study study, it is aimed to perform gingival retraction under rubber-dam isolation by using a 212 clamp (Hu-Friedy, USA), a Brinker B4 clamp (Coltene Hygenic, USA), dental floss using the simple knot tie method, and using the simple knot tie and 212 clamp together. The study was planned as a split mouth. All of these methods will be applied systematically on upper incisors of each patient (teeth numbered 11-12-21-22) by changing them in a clockwise direction. The application time of the retraction methods in each tooth will be limited to 30 minutes, the working time is planned as 2 hours for a total of 4 teeth.

Before starting the treatment, patients will have to sign information and consent forms. In the present study, direct composite restorations are planned under local anesthesia, and it is planned to evaluate the effects of different retraction methods on periodontal tissues and patient comfort. After the retraction technique to be used, direct composite restorations will be performed. Restorations involving the cervical region veneer restorations; It will include aesthetic restorations in the maxillary anterior region, including cervical area. The preparation will only be made when necessary and will protect the hard tissues of the teeth as much as possible in minimally invasive way.

All restorations to be made in our study are planned to be applied with the 'additive' finishing technique. In this technique, the resin material is placed on the tooth surface in small pieces during composite layering and no 'overcontouring' is made. In this way, it is not necessary to reduce the areas close to the gingiva with a drill during the finishing of the restorations, especially concerning the cervical region, and periodontal tissues can be protected. In our study, it is aimed to eliminate the use of burs in the cervical area, which is an important parameter of possible damage to periodontal tissues, and to observe the effects of retraction methods by using this technique.

- Data collection method Changes in periodontal tissues will be evaluate; using plaque index, bleeding on probing, probing depth, keratinized gingiva, attached gingiva, relative gingival margin level, relative attachment level and VAS (visual analogue scale) scoring and patient comfort levels after the procedure at different times (pre-restoration, after restoration). It will be evaluated immediately after, 1 week later, 1 month later, 3 months later. The evaluation time is planned not to exceed 10 minutes, restorations are done by a single specialist in Marmara University Restorative Dentistry Department. Periodontal evaluations will be performed as a single blind, the observer will not know which retraction method is applied to which teeth during the evaluation. Intra-observer agreement will be evaluated, and work will continue in the presence of agreement above 80%.

Restorative materials to be used in the study; Estelite Asteria (Tokuyama, Japan) with nano-hybrid properties will be used as resin composite for the restorations. A 37.5% phosphoric acid (Gel Etchant, Kerr Dental, USA) and a universal agent Tokuyama Universal Bond II (Tokuyama) will be used. For polymerization, Valo Cordless (Ultradent Products, USA) will be used in standard mode (/1000 mw/cm2). In case of, preparation is required, the type of atraumatic burs to be used as much as possible, red or yellow banded diamond burs (Acurata, Japan) and multi-blade tungsten carbide burs (Acurata) will be preferred.

The patients will be isolated with a rubber-dam under local anesthesia and the clamps to be used will be systematically applied to the maxillary incisors.

Nic Tone Thick (Dental Dam, Nic Tone, Romania) will be used as a rubber-dam rubber cover for patients. In addition, sterile frames (Hu-Friedy Group, USA), forceps (Hu-Friedy Group, USA) and puncher (Hu-Friedy Group, USA) will be used as rubber-dam instruments on patients. For gingival retraction, Hu-Friedy #212 clamp (Hu-Friedy Group, USA), Coltene B4 Brinker clamp (Coltene/ Whaledent, Switzerland) and waxed dental floss (gum) will be used.

Clinical Index and Measurements Determination of Gingival Phenotype Evaluating the visibility of the silhouette of the periodontal probe inserted into the sulcus is a technique used to determine the phenotype. If the silhouette of the probe placed in the sulcus is visible, the gingiva is considered thin, and if it is not, the gingiva is considered thick.

Keratinized Gums The distance between the mucogingival junction and the gingival margin will be measured as the width of the keratinized gingiva after the alveolar mucosa is pushed and curved coronally and with periodontal probe and the mucogingival junction is determined.

Attached Gingiva The distance between the mucogingival junction and the floor of gingival sulcus will be measured as the width of the attached gingiva.

Plaque Index For each tooth, plaque index measurements will be made from 4 regions as mesiobuccal, midbuccal, distobuccal, midpalatinal.

Bleeding on Probing Bleeding on probing will be examined in 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal. (+) or (-) values will be given according to the presence or absence of bleeding that occurs after the Unc (University of North Carolina) probe examination.

Probing Depth For each of the initially selected teeth, probing depth measurements will be made in a total of 6 regions: mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.

Visual Analogue Scale (VAS) On the 1st and 7th days after retraction using VAS, the patient will be asked to score the pain in the relevant regions between 1 and 10 according to its severity.

Relative Attachment Level Using the Chu's Gauge handpiece, it will be placed on the incisal edge of the incisors, the incisal guide edge of the handpiece will be taken as the fixed guide point, and the distance between the floor of gingival sulcus and the incisal guide edge will be measured and recorded with a periodontal probe. Relative attachment level measurement will be made in 6 regions, mesiobuccal, midbuccal, distobuccal, mesiopalatinal, midpalatinal, and distopalatinal surfaces of each tooth.

Relative Gingival Margin Level Using the Chu's Gauge handpiece, it will be placed on the incisal edge of the incisors, the incisal guide edge of the handpiece will be taken as the fixed guide point, and the distance between the incisal guide and the gingival margin will be measured and recorded. Relative gingival margin level measurement will be made in a total of 6 regions of each tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual/palatinal, mesiopalatinal, midpalatinal, and distopalatinal surfaces.

Evaluation of Restorations Restorations will be evaluated according to FDI (Fédération Dentaire Internationale) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35
* Have sufficient cognitive ability to understand the consent procedure
* Clinically healthy gingiva and periodontium
* Daily cigarette consumption of 10 or less
* No attachment loss, bleeding on probing, or plaque buildup
* Vital upper teeth (12-22) without signs of irreversible pulpitis
* Patients with cervical lesions, abrasion lesions and/or indications for diastema closure requiring restoration
* Patients with cervical lesions at or below the gingival level
* Patients with direct composite restoration indications concerning the cervical region in their upper anterior 4 incisors.

Exclusion Criteria:

* Any disability (mental health conditions, mentally handicapped and physically handicapped)
* Systemic diseases or serious medical risks (Cardiovascular disorder, diabetes, hypertensive, epileptic)
* Compliance problem, inability to provide post-treatment hygiene
* Gingival hyperplasia or bleeding disorder
* Signs of attachment loss of periodontal disease
* Patients for whom rubber dam placement is contraindicated (patient with asthma diagnosis, mouth breathing, partially erupted tooth, overly malpositioned teeth and latex allergy).
* Signs of periapical pathology or pulpal posterior or anterior pathology
* Non-vital, endodontically treated teeth
* Teeth which have mobility
* Teeth with extraction indication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Relative Attachment Level | Immediately after the restorations
  Relative Attachment Level will measure for the evaluate to effect of different retraction methods on gingival tissue
Relative Attachment Level | 1 week later
  Relative Attachment Level will measure for the evaluate to effect of different retraction methods on gingival tissue
Relative Attachment Level | 1 month later
  Relative Attachment Level will measure for the evaluate to effect of different retraction methods on gingival tissue
Relative Attachment Level | 3 months later
  Relative Attachment Level will measure for the evaluate to effect of different retraction methods on gingival tissue
Relative Gingival Margin Level | Immediately after the restorations
  Relative Gingival Margin Level will measure for the evaluate to effect of different retraction methods on gingival tissue
Relative Gingival Margin Level | 1 week later
  Relative Gingival Margin Level will measure for the evaluate to effect of different retraction methods on gingival tissue
Relative Gingival Margin Level | 1 month later
  Relative Gingival Margin Level will measure for the evaluate to effect of different retraction methods on gingival tissue
Relative Gingival Margin Level | 3 months later
  Relative Gingival Margin Level will measure for the evaluate to effect of different retraction methods on gingival tissue

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Tüter Bayraktar, Asst. Prof, Principal Investigator — Marmara University Faculty of Dentistry
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the article of the study published in an international journal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years
Access Criteria: Data will be shared after the article of the study published in an international journal.